CLINICAL TRIAL: NCT05005689
Title: A Randomised, Controlled Trial to Assess the Effect of Different Modes of Fluoride Delivery on Enamel Demineralisation, During Orthodontic Treatment With Fixed Appliances
Brief Title: Fluoride Delivery to Prevent White Spots During Orthodontic Treatment
Acronym: FL4OWS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5604
Record Dates: First submitted 2021-06-10; First posted 2021-08-13 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Orthodontic Appliance Complication; Tooth Demineralization
Keywords: Fluoride; CPP-ACP
MeSH Terms: conditions — Tooth Demineralization | interventions — Sodium Fluoride; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mouthwash (Active Comparator): Fluoride mouthwash (0.05%; 225ppm) 10ml for 1 minute daily
  Interventions: Drug: Fluoride mouthwash (0.05%; 225ppm).
- Tooth Mousse (Experimental): Tooth Mousse Plus (Recaldent™ CPP-ACP [casein phosphopeptide (CPP)-amorphous calcium phosphate (ACP)] and Sodium Fluoride 0.2% w/w; 900 ppm).
  Tooth creme; 2ml smear daily
  Interventions: Drug: Tooth Mousse Plus

INTERVENTIONS:
Drug: Fluoride mouthwash (0.05%; 225ppm). — Mouthwash
  Other Names: Fluorigard
  Arms: Mouthwash
Drug: Tooth Mousse Plus — Tooth Mousse
  Other Names: Recaldent™ CPP-ACP [casein phosphopeptide (CPP)-amorphous calcium phosphate (ACP)] and Sodium Fluoride 0.2% w/w (900 ppm).
  Arms: Tooth Mousse

SUMMARY:
The aim of this 2-armed, parallel, randomised, controlled trial is to assess the effect of different ways of applying fluoride to teeth on the formation of white spots (enamel demineralisation), during orthodontic treatment with fixed metal braces, in children and adolescents.

DETAILED DESCRIPTION:
One of the most common side-effects and risks of orthodontic treatment with fixed (metal) braces is damage to the outer surface (enamel) of the teeth. This damage can take the form of white or brown spots on the teeth (white spot lesions; WSLs) or if severe, holes in the teeth that need a filling.

The aims of this study are to find out the best way of preventing damage to the teeth of children and adolescents who are under going orthodontic treatment with fixed (metal) braces.

The participants will be 130 children, aged 11-16 years old, inclusive. The participants will be split into two groups using a process called randomisation. The treatments will be standard fluoride toothpaste (Colgate) and either:

1. Fluoride mouth wash (Fluorigard) or
2. Tooth Mousse Plus

The participants' teeth will be checked at every visit and the brace adjusted. Photographs of the participants' teeth will be taken very 3 months to see if any of the teeth have been damaged. The participants will be asked about the impact of their teeth on their life. Participants and parents will be asked about the impact of any white spots that form on the participants' teeth during the treatment with fixed (metal) braces.

The study will follow the participants through the whole length of treatment which will take about 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Planned to receive orthodontic treatment with upper and lower fixed orthodontic appliances (braces) either alone or following a period of functional appliance treatment.
* 11-16 years of age inclusive at the start of the fixed orthodontic appliance treatment.
* All genders.
* Fit and well with no chronic disease necessitating regular hospital follow-up at hospital.
* Willing to participate

Exclusion Criteria:

* Significant disabilities that may affect manual dexterity;
* Any medical complication that would contraindicate the use of the fluoride treatments or milk products;
* Previous orthodontic treatment except Phase I functional appliance treatment;
* From areas that have fluoridated water supply*;
* Full coronal coverage restorations;
* More than 2 missing anterior teeth;
* Showing signs of systemic illness e.g. fever, cough, loss of taste/smell;
* Any abnormality of face, lips e.g. cleft lip and/or palate or craniofacial abnormality or soft tissues of the mouth e.g. aphthous ulcers or connective tissue disorder.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
New white spot lesions (WSLs) | Through to study completion, an average of 2 years
  The incidence of new demineralisation (WSLs), developing on the anterior teeth during fixed orthodontic treatment assessed from white light and quantitative light-induced fluorescence (QLF) images, will be measured.
  Numerical scale 0 - unlikely to be more than 100. Higher score is worse.

SECONDARY OUTCOMES:
Size of white spot lesion (WSL) | Through to study completion, an average of 2 years
  The degree (∆F) of enamel demineralisation on the surfaces of the anterior teeth measure from quantitative light-induced fluorescence (QLF) images.
  Measured as a percentage (%) compared to baseline i.e. loss of mineral. Scale ∆F 0% to -100%; Higher score is worse.
Extent of white spot lesion (WSL) | Through to study completion, an average of 2 years
  The extent (∆Q) of enamel demineralisation on the surfaces of the anterior teeth. measure from quantitative light-induced fluorescence (QLF) images.
  Measured as a percentage per millimetre squared (%mm-2) compared to baseline i.e. loss of mineral. Scale ∆Q 0% to -100%mm-2. Higher score is worse.
Participants' perception of WSL | Through to study completion, an average of 2 years
  Participants' perception of the WSLs. Measured on 100mm visual analogue scale (VAS). Scale 0 to 100. Higher score is worse.
Parents' perception of WSL | Through to study completion, an average of 2 years
  Parents' perception of the WSLs. Measured on 100mm visual analogue scale (VAS). Scale 0 to 100. Higher score is worse.
MIQ Score | Through to study completion, an average of 2 years
  Malocclusion Impact Questionnaire (MIQ) score. Measured using a 17-item questionnaire.
  Total score will be used where minimum score is 0 and maximum score is 34; higher score indicates poorer oral health related quality of life (OHRQoL).

CONTACTS AND LOCATIONS:
Overall Officials: Heather Rogers, Study Chair — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No